CLINICAL TRIAL: NCT05225740
Title: Large-group One-session Exposure Therapy Protocol for Targeting Anxiety Sensitivity
Brief Title: Exposure Therapy Consortium (ETC) for Anxiety Sensitivity
Acronym: ETC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Colorado, Boulder (Other); University of Miami (Other); University of Mississippi, Oxford (Other); Ruhr University of Bochum (Other); Boston University (Other); Fordham University (Other); The University of New South Wales (Other); Southern Methodist University (Other); Institute of Behavioral-Therapy and -Medicine at the Philipps University Marburg (Other); Technische Universität Dresden (Other); Curtin University (Other); Hebrew University of Jerusalem (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Jasper A. Smits, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-09-0153
Record Dates: First submitted 2021-05-17; First posted 2022-02-04 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Elevated Anxiety Sensitivity
Keywords: Exposure Therapy; Harm Expectancy Violation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): General stress reduction based on stress management training to help people cope with feelings of anxiety, used as an active control condition
  Interventions: Behavioral: Stress Management Training
- Standard Exposure (Active Comparator): Psychoeducation about exposure therapy and anxiety sensitivity, interoceptive exposure therapy modeling and practice, and completion of questions about the exercises and the large-group aspect
  Interventions: Behavioral: Standard Exposure
- Enhanced Exposure (Experimental): Psychoeducation about exposure therapy and anxiety sensitivity, interoceptive exposure therapy modeling and practice, and post-exposure processing aimed at emphasizing harm expectancy violation
  Interventions: Behavioral: Enhanced Exposure

INTERVENTIONS:
Behavioral: Standard Exposure — The standard intervention will include an orientation and psychoeducation phase, an exposure practice phase consisting five repeated trials per each of the three exposure exercises, and a post-exposure exercise. The post-exposure exercise will involve completing a set of questions regarding the exercises and the group experience.
  Arms: Standard Exposure
Behavioral: Stress Management Training — Stress management training (SMT) is designed to help people better cope with feelings of anxiety that accompany high levels of anxiety sensitivity. SMT will involve group instruction in healthy ways to experience and cope with stress whenever difficult situations arise. Participants will teach participants ways to maintain a healthy lifestyle, targeting things like nutrition, exercise, and sleep hygiene. This intervention will also involve progressive muscle relaxation training.
  Arms: Control
Behavioral: Enhanced Exposure — The enhanced intervention will include an orientation and psychoeducation phase, an exposure practice phase consisting five repeated trials per each of the three exposure exercises, and a processing exercise. The post-processing exercise will involve completing a set of questions that will highlight harm expectancy violations.
  Arms: Enhanced Exposure

SUMMARY:
The current study seeks to test differences between a single-session large-group format of standard exposure, enhanced exposure, and a control condition in treating anxiety sensitivity. It is hypothesized that 1) participants assigned to either exposure condition will evidence greater reductions in anxiety sensitivity from pre-treatment to posttreatment relative to those in the control condition; 2) participants assigned to the enhanced exposure condition will evidence greater reductions in anxiety sensitivity from pre-treatment to posttreatment relative to those in the standard exposure condition. The investigators will test putative moderators and mechanisms of action. Prior to initiating the study for purposes of data analyses, the investigators will pilot study procedures during Spring 2020.

DETAILED DESCRIPTION:
Anxiety sensitivity (AS), or the fear of anxiety and related sensations, represents an individual difference variable implicated in the risk and maintenance of anxiety and related disorders. Best conceptualized as an amplification factor, AS, when elevated, interacts with changes in bodily sensations (e.g., racing heart, sweating, dizziness) to produce fear. Exposure therapy involves repeated confrontation to feared cues to help individuals reestablish a sense of safety around these cues. Exposure therapy is a transdiagnostic treatment strategy that has shown to be efficacious across anxiety and related disorders. Symptom induction exercises (e.g., spinning, voluntary hyperventilation, straw breathing, using a tongue depressor) are useful for providing exposure to benign bodily sensations (e.g., dizziness, racing heart, breathlessness, choking), allowing individuals with elevated AS to learn that, while perhaps uncomfortable, these sensations are not harmful, but safe.

In an effort to increase the access to exposure therapy, Margraf and colleagues developed a large-group one-session exposure therapy protocols involving brief psychoeducation followed by either observation or participation in exposure practice for fears of various cues, including spiders, dental procedures, and blood, injuries and injections. Initial testing indicates feasibility and shows that individuals participating in these protocols evidence significant improvement in anxiety symptoms.

The current study involves the development and testing of a large-group one-session exposure therapy protocol designed to target AS. The investigators will compare two variants of the protocol and include a general stress reduction protocol as a control condition (CONTROL). The first variant (STANDARD) is a standard protocol, modeled after those developed by Margraf and colleagues, that includes a combination of psychoeducation (about the nature and [exposure] therapy of anxiety sensitivity) and interoceptive exposure therapy modeling and practice. The second variant (ENHANCED) is identical to the first but also includes post-exposure practice processing aimed at facilitating threat reappraisal (i.e., safety learning). All interventions will be delivered in large-group format (N ≥ 25 participants) by a team of clinicians (N = 3) trained in the delivery of exposure therapy. In an effort to improve the quality of research on exposure therapy, another central aim of this study is to examine the feasibility of an exposure therapy consortium. The investigators have established a network of research sites (N=11) with expertise in exposure therapy. With UT as the coordinating site, the investigators propose to implement the study protocol at each of these sites, allowing us to obtain the data needed to examine replication and the identification of predictors, moderators and mediators of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Students currently enrolled in enrolled in an introductory psychology course a psychology course
* Elevated anxiety sensitivity (total ASI-3 score ≥ 23)

Exclusion Criteria:

- History of respiratory or cardiovascular conditions (e.g., asthma, high blood pressure), neurological disorders (e.g., epilepsy), current pregnancy, or medical problems (e.g., inner ear problems, back or joint problems) that may interfere with an ability complete interoceptive exposure procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity | 1 day
  The primary outcome is Anxiety Sensitivity at the posttreatment endpoint. Anxiety Sensitivity will be measured with the Anxiety Sensitivity Index-3 scale (ASI-3; 0-72, lower scores mean better outcome).

SECONDARY OUTCOMES:
Change in Anxiety Sensitivity | 1 month
  Pretreatment to follow-up change in Anxiety Sensitivity as indexed by scores on the Anxiety Sensitivity Index-3 scale (ASI-3; 0-72, lower scores mean better outcome)
Depression | 1 month
  Pretreatment to follow-up change in Depressed Mood as indexed by scores on the Patient Health Questionnaire-8 scale (PHQ-8; 0-24, lower scores mean better outcome)
Anxiety | 1 month
  Pretreatment to follow-up change in Anxiety as indexed by scores on the Generalized Anxiety Disorder-7 scale (GAD-7; 0-21, lower scores mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, PhD, Principal Investigator — The University of Texas at Austin
Locations (12):
- United States (5):
  - The University of Colorado at Boulder, Boulder, Colorado
  - The University of Miami, Miami, Florida
  - Boston University, Boston, Massachusetts
  - The University of Mississippi, Oxford, Mississippi
  - The University of Texas at Austin, Austin, Texas
- Australia (2):
  - University of New South Wales, Kensington
  - Curtin University, Perth
- Germany (4):
  - Philipps-Universität Marburg, Marburg, Hesse
  - Ruhr-Universität Bochum, Bochum, Ruhr Region
  - Technische Universität Dresden, Dresden, Saxony
  - University of Göttingen, Göttingen
- The Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Upon completion of data collection, data from all sites will be pooled and analysis will take place at UT. All data will be encrypted with numeric codes so that no identifying information will be included in analyses. The data, in aggregate form only, may be used for future research or be made available to other researchers for research purposes not detailed in this study.